CLINICAL TRIAL: NCT00800683
Title: Safety in Type 2 Diabetic Patients With Severe Chronic Renal Impairment, 5 mg BI 1356 vs. Placebo, DB, Parallel Group, Randomized, Insulin Background Inclusive
Brief Title: Safety and Efficacy in Type 2 Diabetic Patients With Severe Chronic Renal Impairment, 5 mg BI 1356 (Linagliptin) vs. Placebo, Insulin Background Inclusive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.43; 2008-001569-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- BI 1356 (Experimental): patient to receive a tablet containing BI 1356 once daily
  Interventions: Drug: BI 1356
- placebo (Placebo Comparator): patient to receive a tablet identical to BI 1356 once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: BI 1356 — BI 1356 dosed once daily
  Arms: BI 1356
Drug: placebo — placebo matching BI 1356 taken once daily
  Arms: placebo

SUMMARY:
to determine safety, efficacy and tolerability of BI 1356 versus placebo

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with type 2 diabetes and with glomerular filtration rate (GFR) <30 ml/min, who are not on chronic dialysis.
* Insufficient glycemic control (hemoglobin A1c (HbA1c) between 7.0% and 10.0%)
* Age 18 or over and not older than 80 years

Exclusion criteria:

* Treatment with any other anti diabetic drug other than insulin and/or sulphonylurea within 3 months prior to informed consent
* Myocardial infarction, stroke or transient ischemic attack (TIA) within 6 months prior to informed consent
* Unstable or acute congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- United States (24):
  - 1218.43.10027 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1218.43.10011 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1218.43.10006 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1218.43.10021 Boehringer Ingelheim Investigational Site, Whittier, California
  - 1218.43.10013 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1218.43.10009 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 1218.43.10018 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1218.43.10022 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.43.10015 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1218.43.10016 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1218.43.10003 Boehringer Ingelheim Investigational Site, Great Neck, New York
  - 1218.43.10004 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1218.43.10020 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1218.43.10019 Boehringer Ingelheim Investigational Site, Delaware, Ohio
  - 1218.43.10008 Boehringer Ingelheim Investigational Site, Mentor, Ohio
  - 1218.43.10005 Boehringer Ingelheim Investigational Site, Bethlehem, Pennsylvania
  - 1218.43.10007 Boehringer Ingelheim Investigational Site, Carlisle, Pennsylvania
  - 1218.43.10001 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 1218.43.10025 Boehringer Ingelheim Investigational Site, Aiken, South Carolina
  - 1218.43.10023 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1218.43.10024 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1218.43.10014 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.43.10017 Boehringer Ingelheim Investigational Site, Lufkin, Texas
  - 1218.43.10010 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Australia (7):
  - 1218.43.61009 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1218.43.61010 Boehringer Ingelheim Investigational Site, Auchenflower, Queensland
  - 1218.43.61006 Boehringer Ingelheim Investigational Site, Kippa-Ring, Queensland
  - 1218.43.61007 Boehringer Ingelheim Investigational Site, Reservoir, Victoria
  - 1218.43.61011 Boehringer Ingelheim Investigational Site, Richmond, Victoria
  - 1218.43.61005 Boehringer Ingelheim Investigational Site, Adelaide, SA
  - 1218.43.61002 Boehringer Ingelheim Investigational Site, Herston, QLD
- Hong Kong (2):
  - 1218.43.85201 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1218.43.85203 Boehringer Ingelheim Investigational Site, New Territories
- Israel (9):
  - 1218.43.97008 Boehringer Ingelheim Investigational Site, Afula
  - 1218.43.97005 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1218.43.97003 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.43.97004 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1218.43.97009 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1218.43.97002 Boehringer Ingelheim Investigational Site, Kfar Saba
  - 1218.43.97007 Boehringer Ingelheim Investigational Site, Nahariya
  - 1218.43.97001 Boehringer Ingelheim Investigational Site, Safed
  - 1218.43.97006 Boehringer Ingelheim Investigational Site, Tel Aviv
- New Zealand (4):
  - 1218.43.64001 Boehringer Ingelheim Investigational Site, Auckland
  - 1218.43.64003 Boehringer Ingelheim Investigational Site, Christchurch
  - 1218.43.64004 Boehringer Ingelheim Investigational Site, Takpuna
  - 1218.43.64002 Boehringer Ingelheim Investigational Site, Tauranga
- Ukraine (7):
  - 1218.43.38003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.43.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.43.38006 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.43.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.43.38007 Boehringer Ingelheim Investigational Site, Luhansk
  - 1218.43.38008 Boehringer Ingelheim Investigational Site, Ternopil
  - 1218.43.38002 Boehringer Ingelheim Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] McGill JB, Barnett AH, Lewin AJ, Patel S, Neubacher D, von Eynatten M, Woerle HJ. Linagliptin added to sulphonylurea in uncontrolled type 2 diabetes patients with moderate-to-severe renal impairment. Diab Vasc Dis Res. 2014 Jan;11(1):34-40. doi: 10.1177/1479164113507068. Epub 2013 Oct 29. PMID 24169807

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin (BI 1356): Patients randomized to receive treatment with Linagliptin 5mg
Period: Overall Study
Arm/Group | Placebo | Linagliptin (BI 1356)
Started | 65 (Number who started treatment) | 68 (Number who started treatment)
Completed | 48 (Number who completed treatment) | 49 (Number who completed treatment)
Not Completed | 17 | 19
Not completed — Adverse Event | 11 | 8
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Lack of Efficacy | 1 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin (BI 1356) | Total
Number analyzed (Participants) | 65 | 68 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.6) | 64.0 (10.9) | 64.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 35 | 45 | 80
Glycosylated haemoglobin (HbA1c) at baseline [Mean (Standard Deviation); unit: percentage] — Described in the patients of the Full Analysis Set : 62 in placebo group versus 66 in Linagliptin group
  percentage | 8.2 (0.9) | 8.2 (1.1) | 8.2 (1.0)
Fasting plasma glucose (FPG) at baseline [Mean (Standard Deviation); unit: mg/dL] — Described in the patients of the Full Analysis Set : 62 in placebo group versus 66 in Linagliptin group
  mg/dL | 160.1 (65.4) | 149.5 (79.5) | 154.6 (72.9)
Body Mass Index (BMI) Continuous [Mean (Standard Deviation); unit: kg/m²] | 31.7 (5.9) | 32.3 (5.9) | 32.0 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 12
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline continuous HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set (FAS) included all treated and randomised participants with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | -0.15 (0.15) | -0.76 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); For patients who received rescue medication during the course of the trial, the Oracle Clinical (OC) technique was utilised for all efficacy endpoints and the values were set to missing after the rescue medication was administered; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.60, 95% CI [-0.89 to -0.31], Standard Error of Mean 0.15

2. Secondary Outcome: HbA1c Change From Baseline at Week 52
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 52 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | 0.01 (0.16) | -0.71 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI [-1.03 to -0.41], Standard Error of Mean 0.16

3. Secondary Outcome: HbA1c Change From Baseline at Week 18
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | 0.04 (0.14) | -0.57 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.61, 95% CI [-0.90 to -0.33], Standard Error of Mean 0.14

4. Secondary Outcome: HbA1c Change From Baseline at Week 24
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | 0.04 (0.14) | -0.64 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI [-0.96 to -0.41], Standard Error of Mean 0.14

5. Secondary Outcome: HbA1c Change From Baseline at Week 30
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 30 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | 0.04 (0.16) | -0.67 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI [-1.05 to -0.39], Standard Error of Mean 0.17

6. Secondary Outcome: HbA1c Change From Baseline at Week 36
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 36 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | 0.03 (0.16) | -0.72 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI [-1.06 to -0.44], Standard Error of Mean 0.16

7. Secondary Outcome: HbA1c Change From Baseline at Week 42
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 42 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | -0.08 (0.16) | -0.73 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.64, 95% CI [-0.96 to -0.33], Standard Error of Mean 0.16

8. Secondary Outcome: HbA1c Change From Baseline at Week 48
Description: HbA1c is measured as a Percent. Thus, this change from baseline reflects the Week 48 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for continuous baseline HbA1c , creatinine clearance at baseline and previous anti-diabetic medication.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percent | -0.04 (0.15) | -0.77 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.73, 95% CI [-1.02 to -0.44], Standard Error of Mean 0.15

9. Secondary Outcome: The Occurrence of Treat to Target Efficacy Response, That is an HbA1c Under Treatment of <6.5% After 52 Weeks of Treatment
Description: The percentage of patients with an HbA1c value below 6.5% at week 52 was calculated for each treatment arm. Non-completers were imputed as failure (NCF). Analysis was only performed on patients with baseline HbA1c>=6.5%
Time Frame: Baseline and Week 52
Population: This population includes the FAS with baseline HbA1c>=6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percentage of patients | 0 | 6.1
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.1199, Fisher Exact — P-value calculated using a Fisher's exact Test

10. Secondary Outcome: The Occurrence of a Treat to Target Efficacy Response, That is an HbA1c Under Treatment of <7.0% After 52 Weeks of Treatment
Description: The percentage of patients with an HbA1c value below 7.0% at week 52 was calculated for each treatment arm. Non-completers were imputed as failure (NCF). Analysis was only performed on patients with baseline HbA1c>=7%.
Time Frame: Baseline and Week 52
Population: This population includes the FAS with baseline HbA1c>=7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 61 | 61
Percentage of patients | 9.8 | 18.0
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Linagliptin vs Placebo. The odds-ratio is based on a logistic regression model including baseline HbA1c, previous anti-diabetic medication and creatinine clearance; Test type: Superiority or Other; p = 0.2225, Regression, Logistic; Odds Ratio (OR) = 0.103, 95% CI [0.003 to 3.978]

11. Secondary Outcome: Percentage of Patients With HbA1c Lowering by 0.5% at Week 52
Description: The percentage of patients with an HbA1c reduction from baseline >=0.5% at week 52 was calculated for each treatment arm. Non-completers were imputed as failure (NCF).
Time Frame: Baseline and Week 52
Population: The Full Analysis Set (FAS) included all patients with a baseline and at least one on treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 62 | 66
Percentage of patients | 11.3 | 27.3
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.8927, Regression, Logistic; Odds Ratio (OR) = 0.816, 95% CI 2-sided [0.042 to 15.756]

12. Secondary Outcome: FPG Change From Baseline at Week 12
Description: This change from baseline reflects the week 12 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , creatinine clearance , HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 12
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -7.08 (11.08) | -8.81 (10.66)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.8802, ANCOVA; Mean Difference (Final Values) = -1.73, 95% CI [-24.36 to 20.91], Standard Error of Mean 11.43

13. Secondary Outcome: FPG Change From Baseline at Week 18
Description: Model includes treatment, continuous baseline FPG , creatinine clearance , HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 18
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -12.72 (7.94) | -14.97 (7.64)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.7848, ANCOVA; Mean Difference (Final Values) = -2.24, 95% CI [-18.47 to 13.98], Standard Error of Mean 8.19

14. Secondary Outcome: FPG Change From Baseline at Week 24
Description: This change from baseline reflects the week 24 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , baseline creatinine clearance , baseline HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 24
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -6.22 (7.84) | -16.93 (7.54)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.1878, ANCOVA; Mean Difference (Final Values) = -10.72, 95% CI [-26.74 to 5.31], Standard Error of Mean 8.09

15. Secondary Outcome: FPG Change From Baseline at Week 30
Description: This change from baseline reflects the week 30 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , baseline creatinine clearance , baseline HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 30
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -14.54 (7.68) | -10.12 (7.39)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.5781, ANCOVA; Mean Difference (Final Values) = 4.42, 95% CI [-11.28 to 20.12], Standard Error of Mean 7.92

16. Secondary Outcome: FPG Change From Baseline at Week 36
Description: This change from baseline reflects the week 36 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , baseline creatinine clearance , baseline HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 36
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -11.29 (8.53) | -20.53 (8.20)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.2954, ANCOVA; Mean Difference (Final Values) = -9.24, 95% CI [-26.67 to 8.18], Standard Error of Mean 8.80

17. Secondary Outcome: FPG Change From Baseline at Week 42
Description: This change from baseline reflects the week 42 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , baseline creatinine clearance , baseline HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 42
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -13.25 (8.02) | -8.88 (7.71)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.5984, ANCOVA; Mean Difference (Final Values) = 4.37, 95% CI [-12.02 to 20.75], Standard Error of Mean 8.27

18. Secondary Outcome: FPG Change From Baseline at Week 48
Description: This change from baseline reflects the week 48 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , baseline creatinine clearance , baseline HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 48
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -10.52 (8.26) | -3.45 (7.95)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.4085, ANCOVA; Mean Difference (Final Values) = 7.07, 95% CI [-9.82 to 23.96], Standard Error of Mean 8.53

19. Secondary Outcome: FPG Change From Baseline at week52
Description: This change from baseline reflects the week 52 FPG minus the baseline FPG. Means are treatment adjusted for continuous baseline FPG , baseline creatinine clearance , baseline HbA1c and background of anti diabetic drugs
Time Frame: Baseline and Week 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 57 | 63
mg/dL | -6.81 (7.92) | -5.47 (7.62)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin (BI 1356); Test type: Superiority or Other; p = 0.8698, ANCOVA; Mean Difference (Final Values) = 1.34, 95% CI [-14.84 to 17.52], Standard Error of Mean 8.17

20. Secondary Outcome: Change From Baseline in Antidiabetic Background Therapy Dose at 52 Weeks Compared to Baseline and Over Time
Description: Number of patients with at least one change in daily dose, determined by at least a 10% increase in insulin.
Time Frame: Baseline and Week 52
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 65 | 68
Participants
  Week 1- Week12 | 11 | 17
  Week 12 - Week 52 | 29 | 24
  Overall (Baseline -Week 52) | 33 | 32

21. Secondary Outcome: Clinically Relevant Drug-related Abnormalities for Blood Chemistry, Pulse Rate, Laboratory Parameters and ECG
Description: Clinically relevant drug-related abnormalities for blood chemistry, pulse rate, laboratory parameters and ECG. New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: first administration of randomised treatment to ....
Population: Clinically relevant drug-related abnormalities for blood chemistry, pulse rate, laboratory parameters and ECG
Measure: Number; unit: participants
Arm/Group | Placebo | Linagliptin (BI 1356)
Number analyzed (Participants) | 65 | 68
participants
  Cardiac disorders - Tachycardia | 1 | 0
  Blood amylase increased | 1 | 0
  Blood creatine phosphokinase MB increased | 1 | 1
  Blood creatine phosphokinase increased | 1 | 2
  Glycosylated haemoglobin increased | 0 | 1

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The period of 52 weeks was the maximum of study treatment. Patients were allowed to remain on study medication for up to 52 weeks.
Arm/Group | Placebo | Linagliptin (BI 1356)
Serious Adverse Events (participants affected / at risk) | 27/65 | 25/68
Other Adverse Events (participants affected / at risk) | 50/65 | 61/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Linagliptin (BI 1356) (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 3 | 3
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Parathyroid gland enlargement (Endocrine disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cardiac death (Cardiac disorders) | 1 | 0
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 5
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 3
Urinary retention (Renal and urinary disorders) | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hilar enlargement (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Linagliptin (BI 1356) (N=68)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 3 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 10
Nausea (Gastrointestinal disorders) | 1 | 5
Oedema peripheral (General disorders) | 7 | 7
Bronchitis (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Urinary tract infection (Infections and infestations) | 7 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 2
Blood creatine phosphokinase increased (Investigations) | 7 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 21
Hypoglycaemia (Metabolism and nutrition disorders) | 32 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Headache (Nervous system disorders) | 4 | 2
Renal impairment (Renal and urinary disorders) | 2 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.